CLINICAL TRIAL: NCT07103200
Title: Evaluation of Decision-Making Fatigue After Traumatic Brain Injury (EDIFY)
Brief Title: Evaluation of Decision-Making Fatigue After Traumatic Brain Injury
Acronym: EDIFY
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Minnesota (Other)
Collaborators: Uniformed Services University of the Health Sciences (U.S. Federal Agency); United States Department of Defense (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: IRB-FY2024-887
Record Dates: First submitted 2025-06-25; First posted 2025-08-05 (Actual); Last update posted 2025-08-05 (Actual); Status verified 2025-08

CONDITIONS: TBI (Traumatic Brain Injury)
Keywords: Mild TBI; Decision-Making Fatigue
MeSH Terms: conditions — Brain Injuries, Traumatic

STUDY DESIGN:
Intervention Model Description: Open-label preliminary, prospective cohort
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- COGED (Active Comparator): The COGED task consists of the classic N-back task of working memory-based decision making, followed by a valuation phase. The N-back phase of the task allows calculation of cognitive performance of a working memory task. During valuation, participants receive titrating offers of differing amounts of money to perform different difficulty levels of the N-back. The result is an effort discounting curve used to measure the individual effort cost. Effort discounting curves show the perceived cognitive effort required to complete each level of the task relative to another (typically the 1-back).
  Interventions: Behavioral: COGED
- Restless Bandit (Active Comparator): Participants are presented with three targets (decks of cards) on the screen, which they select with a mouse movement. Each of the three targets is associated with a hidden probability of reward, which drifts unpredictably and independently across trials. This encourages participants to "exploit" good options when they are available, but also occasionally to "explore "other targets, which could become better at any time. Eye Tracking is done at each visit while the participant completes the Restless Bandit tasks.
  Interventions: Behavioral: Restless Bandit

INTERVENTIONS:
Behavioral: COGED — The COGED task consists of the classic N-back task of working memory-based decision making, followed by a valuation phase. The N-back phase of the task allows calculation of cognitive performance of a working memory task. During valuation, participants receive titrating offers of differing amounts of money to perform different difficulty levels of the N-back. The result is an effort discounting curve used to measure the individual effort cost. Effort discounting curves show the perceived cognitive effort required to complete each level of the task relative to another (typically the 1-back).
  Arms: COGED
Behavioral: Restless Bandit — Participants are presented with three targets (decks of cards) on the screen, which they select with a mouse movement. Each of the three targets is associated with a hidden probability of reward, which drifts unpredictably and independently across trials. This encourages participants to "exploit" good options when they are available, but also occasionally to "explore "other targets, which could become better at any time. Eye Tracking is done at each visit while the participant completes the Restless Bandit tasks.
  Arms: Restless Bandit

SUMMARY:
This is a preliminary, prospective, cohort study to investigate the feasibility of using the COGED and Restless Bandit tasks after a mild to moderate traumatic brain injury as well as in healthy controls.

DETAILED DESCRIPTION:
This study aims to measure the effects of traumatic brain injury in the acute and subacute phases of recovery using these two noninvasive computerized assessments (COGED and bandit). All participants engaged in the study will participate in a total of three visits at Hennepin Healthcare Systems, Inc. (HHS). Each visit will consist of surveys and computerized assessments that will help researchers to understand the effects of decision-making on mental fatigue.

ELIGIBILITY:
Inclusion Criteria for TBI Participants:

* Adults 18 years and older
* Diagnosis of a mild to moderate TBI (GCS > 8 on admission)
* Able to perform a computerized assessment
* Willing to attend all scheduled appointments
* Able to undergo the informed consent process

Inclusion Criteria for Healthy Participants:

* Adults 18 years and older
* Able to perform a computerized assessment
* Willing to attend all scheduled appointments
* Able to undergo the informed consent process

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2025-07-01 (Actual); Primary Completion 2029-07-15 (Estimated); Study Completion 2029-07-15 (Estimated)

PRIMARY OUTCOMES:
Feasibility of using COGED and Bandit computerized assessments in evaluating Decision-Making Fatigue after TBI | 4 years
  Feasibility will be calculated using the sum total number of patients who completed at least 80% of study procedures divided by the sum total number of patients, which is a proportion ranging from 0 to 1. We will then determine if that exceeds 0.5, with higher numbers indicating more feasible.

SECONDARY OUTCOMES:
Acceptability of using COGED and Bandit computerized assessments in evaluating Decision-Making Fatigue after TBI | 4 years
  Acceptability will be calculated using the sum total number of patients who liked study procedures divided by the sum total number of patients, which is a proportion ranging from 0 to 1. We will then determine if that exceeds 0.5, with higher numbers indicating more acceptable.

CONTACTS AND LOCATIONS:
Overall Officials: David Darrow, MD, MPH, Principal Investigator — Hennepin Healthcare Research Institute
Locations (1):
- University of Minnesota, Minneapolis, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No